CLINICAL TRIAL: NCT06276959
Title: Comparison of Near-infrared Imaging With Cone Beam Computed Tomography for Proximal Caries Detection in Permanent Dentition: An in Vivo Study.
Brief Title: The Effectiveness of iTero Element 5D NIRI System in Early Proximal Caries Detection in Permanent Teeth
Status: Recruiting | Type: Observational
Sponsor: West China College of Stomatology (Other)
Responsible Party: Principal Investigator, Xia Kai, Attending physician, West China College of Stomatology
Other Study IDs: WCHSIRB-D-2022-430
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The population with a potential risk of proximal caries.
  Interventions: Diagnostic Test: intraoral scanning; Diagnostic Test: clinical oral examination; Diagnostic Test: cone-beam computed tomography

INTERVENTIONS:
Diagnostic Test: intraoral scanning — The patients underwent intraoral scanning using an iTero Element 5D imaging system (Align Technology, San Jose, CA, USA). This imaging system uses near-infrared light with a wavelength of 850 nm and provides multiple layers of data in a single scan, including a three-dimensional (3D) model, two-dimensional (2D) color images, and NIRI mapped to the 3D model
Diagnostic Test: clinical oral examination — Under illumination in the dental unit, a UVE of the proximal surfaces of the patient's entire dentition was conducted by clinicians using a mouth mirror, dental probe, and an air-water syringe. Visual and tactile methods were performed according to the guidelines of the American Dental Association. Clinicians assessed the soundness of the proximal surfaces based on the presence of discoloration, surface alterations, or cavitation.
Diagnostic Test: cone-beam computed tomography — All enrolled patients underwent CBCT scans because clear aligner treatment required real root/bone visualization features. We would like to clarify that due to the retrospective cross-sectional nature of this study, the patients involved were not subjected to radiation beyond what was initially necessary for their orthodontic treatment.

SUMMARY:
As a new emerging technology for the diagnosis of dental caries, near-infrared imaging requires further research and validation to determine its effectiveness. This study aims to compare near-infrared imaging with cone-beam computed tomography (CBCT) to validate the efficiency of near-infrared imaging in diagnosing proximal caries using large-scale clinical data through retrospective cross-sectional studies.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition
* Participants aged 12 and above
* Patients who have undergone iTero Element 5D oral scanning, as well as CBCT imaging, intraoral photography, and clinical oral examination within 1 week
* CBCT or iTero Element 5D oral scanning indicating proximal caries

Exclusion Criteria:

The following teeth were excluded:

* Third molars
* Teeth with gross loss of tooth structure (cavitated carious lesions extending to the occlusal or buccal/lingual surfaces)
* Teeth with amalgam fillings and their adjacent teeth
* Teeth with crown restorations and their adjacent teeth

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent orthodontic treatment at the West China School of Stomatology.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
positive percent agreement | After the interpretation of CBCT, NIRI, and UVE, an average of 10 months.
  Using CBCT as the reference test, positive percent agreement of NIRI, UVE, and a combination of the two index tests in parallel (PAR) for the detection of proximal caries at different depths and in different tooth locations was evaluated.
negative percent agreement | After the interpretation of CBCT, NIRI, and UVE, an average of 10 months.
  Using CBCT as the reference test, negative percent agreement of NIRI, UVE, and a combination of the two index tests in parallel (PAR) for the detection of proximal caries at different depths and in different tooth locations was evaluated.
overall percent agreement | After the interpretation of CBCT, NIRI, and UVE, an average of 10 months.
  Using CBCT as the reference test, overall percent agreement of NIRI, UVE, and a combination of the two index tests in parallel (PAR) for the detection of proximal caries at different depths and in different tooth locations was evaluated.

SECONDARY OUTCOMES:
Proximal caries positive site diagnosed by CBCT | Immediately following CBCT image interpretation.
  Diagnosis of of carious proximal tooth surfaces identified through CBCT. Specifically, the cross-sectional view showing the deepest caries involvement was used for International Caries Detection and Assessment System (ICDAS) scoring and was categorized into shallow caries, moderate caries (ICDAS 1-2), and deep caries (ICDAS 3-6).
Proximal caries positive site diagnosed by near-infrared imaging (NIRI) | Immediately following NIRI image interpretation.
  Owing to the challenges in applying ICDAS scoring for proximal caries detected using NIRI, the classification was either positive (manifest as bright areas) or negative.
Proximal caries positive site diagnosed by unaided visual examination (UVE) | Immediately following clinical oral examination.
  Under illumination in the dental unit, a UVE of the proximal surfaces of the patient's entire dentition was conducted by senior orthodontists using a mouth mirror, dental probe, and an air-water syringe. Visual and tactile methods were performed according to the guidelines of the American Dental Association. Owing to the challenges in applying ICDAS scoring for proximal caries detected using UVE, the classification was either positive (presence of discoloration, surface alterations, or cavitation) or negative.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Stomatology, Sichuan University, Chengdu, Sichuan, China